CLINICAL TRIAL: NCT01424527
Title: Validation of the New COPD Assessment Test Translated Into Korean in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Korean Chronic Obstructive Pulmonary Disease(COPD) Assessment Test Validation Study
Acronym: CAT
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115114
Record Dates: First submitted 2011-07-07; First posted 2011-08-29 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Disease(COPD); COPD Assessment Test(CAT)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — none retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Obstructive Pulmonary Disease: Males and females 40 years of age or older with a diagnosis of COPD

SUMMARY:
This is a cross-sectional validation study, designed to evaluate the discriminative validity of the Chronic Obstructive Pulmonary Disease Assessment Test translated in a local language in patients with Chronic Obstructive Pulmonary Disease.

DETAILED DESCRIPTION:
The Chronic obstructive pulmonary disease Assessment Test is a new questionnaire that has been developed recently to improve communication between doctors and patients. It is known to have good relationship with other measures of quality of life. For the wider application to practice, it has been translated into a local language in many countries.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrolment in the study must meet all of the following criteria:

1. Type of subject: Outpatients
2. Informed consent: Subjects must give their signed and dated written informed consent to participate.
3. Gender: Male or Female
4. Age: 40 years of age or older at a clinic visit
5. COPD diagnosis: Subjects with an established diagnosis of COPD in the past 6 months or before.
6. Tobacco use: Smokers or ex-smokers with a smoking history of more than 10 pack years.

Exclusion Criteria:

1. Asthma: Subjects with a current diagnosis of asthma. Subjects with a prior history of asthma are eligible if COPD is the current diagnosis.
2. Lung diseases: Subjects with current active respiratory disorders other than COPD, e.g. lung cancer, tuberculosis.
3. Non-compliance: Unable to complete questionnaires

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females 40 years of age or older with a diagnosis of COPD are eligible. Subjects will complete questionnaires and perform spirometry at a single visit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient of the Chronic obstructive pulmonary disease Assessment Test with St George's Respiratory Questionnaire | 1 day
  Correlation coefficient of the Chronic obstructive pulmonary disease Assessment Test with St George's Respiratory Questionnaire

SECONDARY OUTCOMES:
Correlation coefficient of the Chronic obstructive pulmonary disease Assessment Test with Medical Research Council Dyspnea Index | 1 day
  Correlation coefficient of the Chronic obstructive pulmonary disease Assessment Test with Medical Research Council Dyspnea Index
Correlation coefficient of the Chronic obstructive pulmonary disease Assessment Test with Forced expiratory volume in 1 second value. | 1 day
  Correlation coefficient of the Chronic obstructive pulmonary disease Assessment Test with Forced expiratory volume in 1 second

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; Jung, Principal Investigator — Hallym University Medical Center
Locations (5):
- South Korea (5):
  - GSK Investigational Site, Anyang-si
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Gyung Gi Do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul